CLINICAL TRIAL: NCT00336479
Title: A Phase 2 Study of VX-950 in Combination With Peginterferon Alfa-2a (Pegasys®), With Ribavirin (Copegus®) in Subjects With Genotype 1 Hepatitis C Who Have Not Received Prior Treatment
Brief Title: Phase 2 Study of VX-950, Pegasys®, and Copegus® in Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX05-950-104
Record Dates: First submitted 2006-06-09; First posted 2006-06-13 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — telaprevir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week (Placebo Comparator): Placebo (PBO) matched to telaprevir tablet orally thrice daily for 12 weeks in combination with pegylated interferon alfa 2a (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (RBV) tablet orally twice daily at a dose of 1000 milligram per day (mg/day) for subjects weighing less than (<) 75 kilogram (kg) and 1200 mg/day for subjects weighing greater than or equal to (>=) 75 kg, for 48 weeks.
  Interventions: Drug: Ribavirin; Drug: Pegylated Interferon Alfa 2a; Other: Placebo
- Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week (Experimental): Single loading dose of telaprevir 1250 mg tablet orally on Day 1 followed by 750 mg telaprevir tablet thrice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 48 weeks.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Drug: Pegylated Interferon Alfa 2a
- Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week (Experimental): Single loading dose of telaprevir 1250 mg tablet orally on Day 1 followed by 750 mg telaprevir tablet thrice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 24 weeks.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Drug: Pegylated Interferon Alfa 2a
- Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week (Experimental): Single loading dose of telaprevir 1250 mg tablet orally on Day 1 followed by 750 mg telaprevir tablet thrice daily in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 12 weeks.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Drug: Pegylated Interferon Alfa 2a

INTERVENTIONS:
Drug: Telaprevir — tablet
  Other Names: VX-950
  Arms: Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week; Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week; Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week
Drug: Ribavirin — tablet
  Other Names: RBV
Drug: Pegylated Interferon Alfa 2a — Solution for injection
  Other Names: Peg-IFN-alfa-2a
Other: Placebo — matching placebo tablet
  Arms: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week

SUMMARY:
Study the effectiveness of telaprevir (VX-950) in combination with Pegylated Interferon Alfa 2a (Peg-IFN-alfa-2a) and Ribavirin (RBV) in reducing plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C virus Genotype 1 with detectable plasma hepatitis C virus RNA
* Have been infected with hepatitis C virus for greater than (>) 6 months
* Seronegative for hepatitis B surface antigen and Human Immunodeficiency Virus 1 and 2
* Must agree to use 2 methods of contraception, including 1 barrier method, during and for 24 weeks after the completion of the study (unless the subject is a female of documented non-child-bearing potential)
* Female subjects must have a negative pregnancy test at all visits before the first dose

Exclusion Criteria:

* Received any approved or investigational drug or drug regimen for the treatment of hepatitis C
* Any medical contraindications to Pegylated Interferon Alfa 2a or Ribavirin therapy
* Any other cause of significant liver disease in addition to hepatitis C; this may include but is not limited to, hepatitis B, drug or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, Nonalcoholic Steatohepatitis or primary biliary cirrhosis
* Diagnosed or suspected hepatocellular carcinoma
* Histologic evidence of hepatic cirrhosis (including compensated cirrhosis) based on a liver biopsy taken within 2 years before study start
* Alcohol abuse or excessive use in the last 12 months
* Participation in any investigational drug study within 90 days before drug administration or participation in more than 2 drug studies in the last 12 months (exclusive of the current study)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2006-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (37):
- United States (36):
  - Call For Information, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University Liver Research, Palo Alto, California
  - Call For Information, San Francisco, California
  - University of Colorado Hospital, Denver, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Shands Hospital University of Florida, Gainesville, Florida
  - Call for Information, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Clarian Hospital, Indianapolis, Indiana
  - Gulf Coast Research Associates, Baton Rouge, Louisiana
  - Call For Information, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Call for Information, Boston, Massachusetts
  - Call For Information, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Call For Information, Rochester, Minnesota
  - Saint Louis University, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Call For Information, Manhasset, New York
  - Call for Information, New York, New York
  - Columbia University Medical Center, New York, New York
  - Call For Information, Chapel Hill, North Carolina
  - Call For Information, Durham, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Fox Chase/ Temple Cancer Center, Philadelphia, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Methodist Hospital of Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Inova Fairfax Hospital, Annandale, Virginia
  - University of Virginia Health System, Charlotteville, Virginia
  - Metropolitan Research, Fairfax, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico

REFERENCES:
- [Derived] McHutchison JG, Everson GT, Gordon SC, Jacobson IM, Sulkowski M, Kauffman R, McNair L, Alam J, Muir AJ; PROVE1 Study Team. Telaprevir with peginterferon and ribavirin for chronic HCV genotype 1 infection. N Engl J Med. 2009 Apr 30;360(18):1827-38. doi: 10.1056/NEJMoa0806104. PMID 19403902

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 263 subjects were enrolled, of which 13 subjects discontinued the study prior to study drug administration. A total of 250 subjects started treatment.
Period: Overall Study
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week
Started | 75 | 79 | 79 | 17
Completed | 38 | 54 | 53 | 13
Not Completed | 37 | 25 | 26 | 4
Not completed — Adverse Event | 8 | 11 | 18 | 4
Not completed — Noncompliant | 1 | 7 | 3 | 0
Not completed — Physician Decision | 2 | 3 | 1 | 0
Not completed — Lost to Follow-up | 3 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 3 | 0
Not completed — Other | 0 | 0 | 1 | 0
Not completed — Virologic Stopping Rule | 20 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis set included all randomized subjects who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week | Total
Number analyzed (Participants) | 75 | 79 | 79 | 17 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 75 | 79 | 79 | 17 | 250
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (8.7) | 48.7 (7.4) | 48.4 (7.6) | 49.1 (8.0) | 48.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 25 | 5 | 93
  Male | 43 | 48 | 54 | 12 | 157
Region of Enrollment [Number; unit: participants]
  North America | 75 | 79 | 79 | 17 | 250

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Undetectable Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Week 24 After the Completion of Study Drug Dosing
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of detection was 10 international units per milliliter (IU/mL).
Time Frame: 24 weeks after the completion of study drug dosing (up to Week 72)
Population: The Full Analysis set included all randomized subjects who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week
Number analyzed (Participants) | 75 | 79 | 79 | 17
percentage of participants | 41.3 [30 to 53] | 67.1 [56 to 77] | 60.8 [49 to 72] | 35.3 [14 to 62]
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week; Test type: Superiority or Other; p = 0.0014, Regression, Logistic; Treatment, weight, race and baseline HCV RNA as factors; Odds Ratio (OR) = 2.985, 95% CI 2-sided [1.525 to 5.842]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week; Test type: Superiority or Other; p = 0.0204, Regression, Logistic; Odds Ratio (OR) = 2.170, 95% CI 2-sided [1.127 to 4.178]

2. Secondary Outcome: Percentage of Subjects With Undetectable Plasma HCV RNA at Week 12 After the Completion of Study Drug Dosing
Description: as for outcome 1
Time Frame: 12 weeks after the completion of study drug dosing (up to Week 60)
Population: The Full Analysis set included all randomized subjects who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week
Number analyzed (Participants) | 75 | 79 | 79 | 17
percentage of participants | 36.0 [25 to 48] | 58.2 [47 to 69] | 53.2 [42 to 64] | 35.3 [14 to 62]
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week; Test type: Superiority or Other; p = 0.0051, Regression, Logistic; Odds Ratio (OR) = 2.586, 95% CI 2-sided [1.331 to 5.025]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week; Test type: Superiority or Other; p = 0.0418, Regression, Logistic; Odds Ratio (OR) = 1.976, 95% CI 2-sided [1.026 to 3.807]

3. Secondary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any adverse change from the subject's baseline (pre-treatment) condition, including any adverse experience, abnormal recording or clinical laboratory assessment value which occurs during the course of the study, whether it is considered related to the study drug or not. An adverse event includes any newly occurring event or previous condition that has increased in severity or frequency since the administration of study drug. SAE: medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. "Study drug" includes all investigational agents (including placebo, if applicable) administered during the course of the study.
Time Frame: Baseline up to Week 48
Population: The Full Analysis set included all randomized subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week
Number analyzed (Participants) | 75 | 79 | 79 | 17
participants
  AEs | 75 | 79 | 79 | 17
  SAEs | 4 | 5 | 10 | 3

4. Secondary Outcome: Number of Subjects With Viral Relapse
Description: Viral relapse was defined as having detectable HCV RNA during antiviral follow-up. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of detection was 10 international units per milliliter (IU/mL).
Time Frame: After last dose of study drug up to antiviral follow-up (up to Week 72)
Population: Analysis population included subjects who completed their assigned study drug treatment and had undetectable HCV RNA at the completion of treatment (up to Week 48).
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week
Number analyzed (Participants) | 35 | 51 | 41 | 9
participants | 8 | 3 | 1 | 3

5. Secondary Outcome: Maximum (Cmax), Minimum (Cmin) and Average (Cavg) Plasma Concentration of Telaprevir
Description: Only subjects who received telaprevir were to be analyzed for this outcome. Maximum, minimum and average plasma concentrations observed during assessment period were reported.
Time Frame: Day 1, 4, 8, 15, 22, 29, 43, 57, 71, 85
Population: Pharmacokinetic population included all subjects who provided pharmacokinetic assessments and had evaluable and interpretable data.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Telaprevir: All Subjects from "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week", "Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week", and "Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week" reporting groups who received single loading dose of telaprevir 1250 mg tablet orally on Day 1 followed by 750 mg telaprevir tablet thrice daily for 12 weeks.
Arm/Group | Telaprevir
Number analyzed (Participants) | 175
nanogram per milliliter (ng/mL)
  Cmax | 3032.48 (756.93)
  Cmin | 2235.51 (618.37)
  Cavg | 2738.46 (699.06)

ADVERSE EVENTS:
Time Frame: AEs and SAEs During Dosing From Baseline to Week 48
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week
Serious Adverse Events (participants affected / at risk) | 4/75 | 5/79 | 10/79 | 3/17
Other Adverse Events (participants affected / at risk) | 75/75 | 79/79 | 79/79 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week (N=75) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week (N=79) | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week (N=79) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week (N=17)
BRONCHITIS BACTERIAL (Infections and infestations) | 0 | 1 | 0 | 0
FURUNCLE (Infections and infestations) | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 1
LOBAR PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
LYMPHADENITIS (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0 | 0 | 0
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
SCOTOMA (Eye disorders) | 0 | 1 | 0 | 1
RETINAL EXUDATES (Eye disorders) | 0 | 0 | 0 | 1
RETINAL INFARCTION (Eye disorders) | 0 | 1 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1 | 0
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
ADRENAL DISORDER (Endocrine disorders) | 0 | 0 | 1 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 0 | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 1 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
LUMBAR RADICULOPATHY (Nervous system disorders) | 0 | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week (N=75) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 48 Week (N=79) | Telaprevir 12 Week +Peg-IFN-alfa-2a,RBV 24 Week (N=79) | Telaprevir 12 Week+Peg-IFN-alfa-2a,RBV 12 Week (N=17)
FATIGUE (General disorders) | 57 | 58 | 55 | 14
INFLUENZA LIKE ILLNESS (General disorders) | 32 | 30 | 39 | 6
INJECTION SITE ERYTHEMA (General disorders) | 18 | 25 | 22 | 6
PYREXIA (General disorders) | 22 | 15 | 16 | 2
IRRITABILITY (General disorders) | 22 | 8 | 13 | 2
CHILLS (General disorders) | 14 | 18 | 8 | 3
PAIN (General disorders) | 15 | 6 | 9 | 1
PHARMACEUTICAL PRODUCT COMPLAINT (General disorders) | 2 | 8 | 4 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 2 | 1 | 5 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 3 | 4 | 0
FEELING HOT (General disorders) | 0 | 4 | 2 | 0
MALAISE (General disorders) | 1 | 0 | 2 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 17 | 32 | 38 | 4
RASH (Skin and subcutaneous tissue disorders) | 20 | 32 | 24 | 6
DRY SKIN (Skin and subcutaneous tissue disorders) | 19 | 13 | 14 | 1
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 4 | 9 | 18 | 3
ALOPECIA (Skin and subcutaneous tissue disorders) | 8 | 13 | 8 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 14 | 8 | 3
HYPOTRICHOSIS (Skin and subcutaneous tissue disorders) | 7 | 8 | 6 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 3 | 6 | 4 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 8 | 4 | 1 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 3 | 2 | 6 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 3
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 3 | 4 | 2 | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 2 | 3 | 5 | 0
INCREASED TENDENCY TO BRUISE (Skin and subcutaneous tissue disorders) | 2 | 3 | 3 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 3 | 4 | 2 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 2 | 2 | 4 | 0
ECZEMA ASTEATOTIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 22 | 38 | 44 | 11
DIARRHOEA (Gastrointestinal disorders) | 21 | 27 | 33 | 4
VOMITING (Gastrointestinal disorders) | 9 | 16 | 19 | 3
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 13 | 10 | 4
DYSPEPSIA (Gastrointestinal disorders) | 7 | 8 | 7 | 1
DRY MOUTH (Gastrointestinal disorders) | 5 | 8 | 8 | 1
CONSTIPATION (Gastrointestinal disorders) | 4 | 8 | 6 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 | 4 | 6 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 3 | 6 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 6 | 1 | 5 | 2
FLATULENCE (Gastrointestinal disorders) | 3 | 6 | 3 | 1
ANAL DISCOMFORT (Gastrointestinal disorders) | 2 | 3 | 6 | 1
STOMACH DISCOMFORT (Gastrointestinal disorders) | 6 | 1 | 4 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4 | 2 | 4 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 5 | 4 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 3 | 2 | 2 | 1
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 2 | 2 | 4 | 0
PAINFUL DEFAECATION (Gastrointestinal disorders) | 0 | 1 | 4 | 1
PRURITUS ANI (Gastrointestinal disorders) | 0 | 1 | 4 | 1
CHAPPED LIPS (Gastrointestinal disorders) | 2 | 1 | 1 | 1
GINGIVAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 1
LOOSE TOOTH (Gastrointestinal disorders) | 0 | 0 | 0 | 1
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 45 | 34 | 37 | 9
DIZZINESS (Nervous system disorders) | 14 | 15 | 22 | 4
DYSGEUSIA (Nervous system disorders) | 8 | 8 | 8 | 0
DISTURBANCE IN ATTENTION (Nervous system disorders) | 7 | 6 | 4 | 3
MEMORY IMPAIRMENT (Nervous system disorders) | 7 | 2 | 7 | 0
TREMOR (Nervous system disorders) | 1 | 3 | 3 | 1
HYPOAESTHESIA (Nervous system disorders) | 1 | 1 | 4 | 1
HYPERAESTHESIA (Nervous system disorders) | 0 | 4 | 2 | 0
PARAESTHESIA (Nervous system disorders) | 2 | 1 | 2 | 1
SOMNOLENCE (Nervous system disorders) | 1 | 1 | 0 | 2
PAROSMIA (Nervous system disorders) | 2 | 0 | 0 | 1
POOR QUALITY SLEEP (Nervous system disorders) | 1 | 0 | 0 | 1
COGNITIVE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 1
MENTAL IMPAIRMENT (Nervous system disorders) | 0 | 0 | 0 | 1
TENSION HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 1
INSOMNIA (Psychiatric disorders) | 29 | 27 | 35 | 6
DEPRESSION (Psychiatric disorders) | 13 | 15 | 17 | 2
ANXIETY (Psychiatric disorders) | 13 | 11 | 6 | 3
MOOD SWINGS (Psychiatric disorders) | 3 | 5 | 2 | 1
LIBIDO DECREASED (Psychiatric disorders) | 2 | 4 | 1 | 0
TEARFULNESS (Psychiatric disorders) | 0 | 2 | 1 | 1
AGITATION (Psychiatric disorders) | 0 | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 16 | 17 | 13 | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 18 | 15 | 9 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 | 8 | 6 | 2
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 | 7 | 8 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 7 | 4 | 4 | 2
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 | 16 | 17 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 12 | 3
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 4 | 3
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 5 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 5 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 2 | 0
ANAEMIA (Blood and lymphatic system disorders) | 20 | 23 | 29 | 6
NEUTROPENIA (Blood and lymphatic system disorders) | 18 | 19 | 11 | 0
SINUSITIS (Infections and infestations) | 7 | 4 | 4 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 6 | 5 | 0
NASOPHARYNGITIS (Infections and infestations) | 4 | 2 | 2 | 1
CELLULITIS (Infections and infestations) | 0 | 2 | 2 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 1 | 0 | 1
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 0 | 1
VISION BLURRED (Eye disorders) | 6 | 14 | 10 | 3
DRY EYE (Eye disorders) | 3 | 3 | 4 | 1
PHOTOPHOBIA (Eye disorders) | 1 | 4 | 1 | 1
CONJUNCTIVITIS (Eye disorders) | 1 | 0 | 1 | 2
EYE PRURITUS (Eye disorders) | 2 | 0 | 0 | 1
VITREOUS FLOATERS (Eye disorders) | 0 | 2 | 0 | 1
LACRIMATION INCREASED (Eye disorders) | 0 | 1 | 0 | 1
OCULAR ICTERUS (Eye disorders) | 1 | 0 | 0 | 1
SCOTOMA (Eye disorders) | 0 | 1 | 0 | 1
CATARACT (Eye disorders) | 0 | 0 | 0 | 1
RETINAL EXUDATES (Eye disorders) | 0 | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 9 | 11 | 10 | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 | 3 | 4 | 0
ANOREXIA (Metabolism and nutrition disorders) | 4 | 0 | 2 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 5 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
HAEMOGLOBIN DECREASED (Investigations) | 2 | 4 | 4 | 1
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0 | 2 | 1
WEIGHT DECREASED (Investigations) | 0 | 1 | 0 | 1
TINNITUS (Ear and labyrinth disorders) | 4 | 0 | 6 | 0
VERTIGO (Ear and labyrinth disorders) | 2 | 2 | 2 | 1
POLLAKIURIA (Renal and urinary disorders) | 2 | 3 | 5 | 0
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
CONTACT LENS COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
FLUSHING (Vascular disorders) | 1 | 0 | 1 | 1
PALPITATIONS (Cardiac disorders) | 3 | 2 | 0 | 1
JAUNDICE (Hepatobiliary disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days